CLINICAL TRIAL: NCT07100457
Title: Association of OR6A2 Expression on Monocytes With Inflammation and Major Adverse Cardiovascular Events in Myocardial Ischemia-Reperfusion Injury
Brief Title: OR6A2 on Monocytes and Cardiovascular Outcomes in Myocardial Ischemia-Reperfusion Injury
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Genshan Ma, Director of Cardiovascular Medicine & Deputy Director of Cardiovascular Disease Research Institute, Zhongda Hospital Southeast University; Professor (Level-II); Chief Physician; PhD Advisor; Chairman, Cardiovascular Society of Jiangsu Medical Association, Southeast University, China
Other Study IDs: 2020ZDSYLL051-P01
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Ischemia-Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 44 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Myocardial Ischemia-Reperfusion Injury
  Interventions: Diagnostic Test: Blood Biomarker Profiling and Prognostic Follow-up

INTERVENTIONS:
Diagnostic Test: Blood Biomarker Profiling and Prognostic Follow-up — Peripheral venous blood collection for in-vitro quantification of serum biomarkers (including octanal, OR6A2, and inflammatory mediators) via mass spectrometry/ELISA/flow cytometry, coupled with longitudinal surveillance of Major Adverse Cardiovascular Events (MACEs) using hospital records, patient interviews, and adjudicated endpoint verification during scheduled follow-up visits.

SUMMARY:
This study examines how the interaction between octanal (an OR6A2 receptor activator) and OR6A2 expression influences inflammation and clinical outcomes in Myocardial Ischemia-Reperfusion Injury patients. We analyze two key relationships: 1) The octanal-OR6A2 pathway's association with systemic oxidative stress/inflammatory biomarkers, and 2) How OR6A2 expression patterns on monocyte subtypes and plasma octanal levels correlate with major cardiovascular events. Patients undergoing this post-revascularization injury provided blood samples for OR6A2/octanal/inflammation measurements. IR Injury patients underwent 44-month clinical follow-up. Results may identify biological markers for personalized risk assessment after revascularization therapies. Ethics approval: Zhongda Hospital #2020ZDSYLL051-P01.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myocardial infarction (AMI) patients with angiographically-confirmed coronary artery disease undergoing primary percutaneous coronary intervention (PCI), and subsequently diagnosed with protocol-defined myocardial ischemia-reperfusion injury during the post-PCI period.
2. Age 18-90 years inclusive.

Exclusion Criteria:

1. Active systemic infections.
2. Advanced heart failure (NYHA class III-IV).
3. Acute cerebrovascular conditions.
4. Active myocarditis.
5. cardiomyopathy.
6. Refractory ventricular tachycardia/fibrillation.
7. Diagnosis/concurrent treatment for malignancy within 5 years (except non-melanoma skin cancer/carcinoma in situ).
8. Severe renal insufficiency (estimated glomerular filtration rate [eGFR] <30 mL/min/1.73m2 or dialysis dependence).
9. Child-Pugh class C hepatic dysfunction.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutively enrolled participants with myocardial ischemia-reperfusion injury who are recruited from the Department of Cardiology at Zhongda Hospital, Southeast University, China.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | From enrollment to 44 months after reperfusion injury
  Major Adverse Cardiovascular Events (MACEs) defined as the composite endpoint of recurrent acute myocardial infarction, cardiac death, stroke, hospitalization for unstable angina, or unplanned coronary revascularization.

SECONDARY OUTCOMES:
Serum IL-1α Level | Baseline (within 24 hours after confirmed myocardial ischemia-reperfusion injury)
  Units: pg/mL
Serum IL-1β Level | Baseline (within 24 hours after confirmed myocardial ischemia-reperfusion injury)
  Units: pg/mL
Plasma Malondialdehyde (MDA) Level | Baseline (within 24 hours after confirmed myocardial ischemia-reperfusion injury)
  Units: μmol/L
Plasma Hydrogen Peroxide (H₂O₂) Level | Baseline (within 24 hours after confirmed myocardial ischemia-reperfusion injury)
  Units: μmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT07100457/Prot_SAP_000.pdf